CLINICAL TRIAL: NCT07263321
Title: Optimising Treatment for Patients With Depressive Episodes in General Practice Through Algorithm-Based Treatment: A Randomised, Open-label Controlled Trial.
Brief Title: Improving Treatment for Depression in General Practice Using a Step-by-Step Care Plan.
Acronym: ODEGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, René Ernst Nielsen, MD, Professor and PhD., Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20250019
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorder; Depression - Major Depressive Disorder; Depressive Disorder, Major Depressive Disorder; Depressive Disorders; Depression; Depressive Episodes; Depressive Episode
Keywords: Treatment for depressive disorder in General Practice; Algorithm-based treatment in General Practice; Algorithm-guided treatment in General Practice; Algorithm-based treatment for depression in General Practice; Algorithm-based treatment for depressive disorder in General Practice; Algorithm-based treatment for depressive episodes in General Practice; Algorithm-guided treatment for depressive episodes in General Practice; Optimising treatment for depressive episodes in general practice
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual by a general practitioner (TAU-GP). (Other): The participants in this arm will receive "treatment as usual" (TAU), administered by a general practitioner (GP), i.e. the practitioner will implement a standard treatment (e.g. pharmacological) that he or she would normally use when treating a patient with depression in general practice.
  Interventions: Other: Treatment as usual (TAU)
- Treatment as usual by a psychologist (TAU-P). (Other): The participants in this arm will receive "treatment as usual", meaning a standard treatment in the form of Cognitive Behavioural Therapy (CBT) administered by a psychologist (P).
  Interventions: Other: Treatment as usual (TAU)
- Algorithm-based pharmacological treatment by a general practitioner (ALGO). (Experimental): In this arm the general practitioner designs a pharmacological, pre-determined and structured step-by-step care plan, including measurement-based care (e.g. Hamilton Rating Scale for Depression), critical decision points and follow ups at week 4, 8 and 12. At these decision points, rating scales are reviewed, and the score results will trigger the next action according to the pre-determined plan.
  Interventions: Other: Algorithm-Based Treatment

INTERVENTIONS:
Other: Algorithm-Based Treatment — This is an open-label pharmacological intervention.
  Other Names: ALGO; Algorithm-guided treatment; Algorithm treatment
  Arms: Algorithm-based pharmacological treatment by a general practitioner (ALGO).
Other: Treatment as usual (TAU) — This is a "treatment as usual" provided by a general practitioner (GP). The GP will implement a standard treatment he or she normally would use, when treating a patient with moderate depression in general practice.
  Other Names: Treatment as usual by a general practitioner; TAU-GP
  Arms: Treatment as usual by a general practitioner (TAU-GP).
Other: Treatment as usual (TAU) — This is a "treatment as usual" provided by a psychologist (P). The psychologist will implement Cognitive Behavioural Therapy as the standard treatment, since this is a widely used and recognised treatment strategy for patients with depression.
  Other Names: Treatment as usual by a psychologist; TAU-P
  Arms: Treatment as usual by a psychologist (TAU-P).

SUMMARY:
The goal of this clinical trial is to compare three different treatments for depression in patients with moderate depression in General Practice, aged 18-65 years.

We wish to investigate the effect of the treatment approaches, and 171 patients will be included in the trial. The participants will be randomised to one of the following three treatments:

1. Standard treatment provided by a general practitioner (i.e. the general practitioner treats the patient as he/she would normally do, when treating a patient with depression).
2. Standard treatment provided by a psychologist in the form behavioural therapy (i.e. the psychologist treats the patient as he/she would normally do, when treating a patient with depression).
3. A step-by-step treatment plan carried out by a general practitioner. The plan includes pre-determined follow-ups and a pre-determined, structured plan for which medications to use and when to increase dose or switch medication.

The hypothesis is that a structured and step-by-step treatment approach regarding patients with depression, treated in general practice, is more effective than standard treatment provided by a general practitioner and a psychologist.

All the participants will:

1. Receive one of the three treatments for 12 weeks.
2. Have meetings with the project staff every 4 weeks (week 0, 4, 8 and 12) were rating scales will be completed, e.g. a rating scale to measure progress or deterioration in the participant's depression.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be referred to the study with a diagnosis of unipolar depressive disorder, as judge by the GP.
2. Severity of the depressive episode corresponding to moderate depression, as judged by the GP.
3. Clinical uncertainty regarding which of the treatments, medication or psychotherapy, would be the better choice in the case concerned.
4. Age criteria: Participants must be at least 18 years old and no more than 65 years old at the time of randomisation.
5. The participant must be a patient in general practice.
6. Participants must be able to participate in virtual meetings (e.g. by phone or computer) and have e-Boks.
7. The participant must be willing to receive psychotherapy by a psychologist and/or medication.
8. Must have signed the document of informed consent.

Exclusion Criteria:

1. Misuse of substances that might influence the study, as judged by the investigator.
2. Difficulty in understanding the Danish language, as judged by the investigator.
3. A diagnosis of dementia.
4. Medical conditions that might interfere with the study outcome or safety, judged so by the investigator.
5. Pregnancy.
6. High risk of non-adherence at the investigator's discretion.
7. Suicidality: according to C-SSRS with a positive response to question 4 or 5 within the last three months or upon investigator's discretion.
8. No current medical or psychotherapy treatment initiated within the last 4 weeks prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The Hamilton Rating Scale for Depression, 6 item version (HAM-D6) | From enrollment to the end of treatment at 12 weeks.

SECONDARY OUTCOMES:
The Columbia-Suicide Severity Rating Scale (C-SSRS) | From enrollment to the end of treatment at 12 weeks.
The Major Depression Inventory (MDI) | From enrollment to the end of treatment at 12 weeks.
The Personal and Social Performance Scale (PSP) | From enrollment to the end of treatment at 12 weeks
The Danish Adult Reading Test (DART) | At enrollment
The Brief INSPIRE-O | At the end of the treatment at 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Department of Psychiatry, Aalborg, Denmark

DOCUMENTS (1):
  • Study Protocol (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT07263321/Prot_000.pdf